CLINICAL TRIAL: NCT01868295
Title: The Effect of Nocturnal Wear of Dentures on Sleep and Oral Health Related Quality of Life: a Randomized Cross-Over Trial
Brief Title: The Effect of Nocturnal Wear of Dentures on Sleep and Oral Health Related Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Elham Emami, Professor, Université de Montréal
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMD-UdeM-EE-2013a
Record Dates: First submitted 2013-05-29; First posted 2013-06-04 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Sleep; Dentures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sleeping with denture (Experimental): Sleeping with denture at night
  Interventions: Behavioral: Sleeping with denture
- Sleeping without denture (No Intervention): Sleeping without denture at night

INTERVENTIONS:
Behavioral: Sleeping with denture — Sleeping with denture at night
  Arms: Sleeping with denture

SUMMARY:
Tooth loss and sleep problems are common conditions in elders. Tooth loss can influence sleep quality by changing the shape of the lower face and upper airway. While some studies suggest that sleeping without dentures can worsen sleep quality in toothless elders, others suggest the opposite. Consequently, there are currently no evidence-based practice guidelines regarding whether dentures should be used at night, and dentists and doctors do not know how to properly advise their patients on these issues. To address this knowledge gap, over the past 5 years we have carried out research examining the quality of sleep of a group of edentulous elders. In addition, we conducted a pilot study to examine the link between night-time denture wear and sleep. Our results indicate that edentulous elders who wore their dentures at night had high levels of daytime sleepiness. Furthermore, use of dentures at night seemed to increase the risk of apneic events in those elders who had mild sleep disturbance. While intriguing, these results require confirmation in larger samples. In line with our previous research, the aim of the proposed study is to produce reliable evidence that clinical practice guidelines could be based on and which could be used by dentists and doctors who treat toothless elders.

We will enroll 70 toothless elders who will be randomly assigned to wear and not wear their dentures at night for two periods of 30 days. Sleep studies will be conducted at the homes of participants. The participants will also be asked to respond to questions on sleep quality and oral health-related quality of life. Ultimately, the results of this study will help improve the health and quality of life of millions of elders in Canada and around the world.

DETAILED DESCRIPTION:
BACKGROUND

Aging substantially increases the risk of edentulism and sleep disturbance. These two chronic conditions have serious adverse consequences for the functioning and quality of life of elders and place a significant burden on the Canadian health care system. Edentulism can disturb sleep through the alteration of the craniofacial structure and surrounding soft tissue. However, the effect of prosthetic rehabilitation of edentulism on sleep quality is still not well understood. While there is some evidence suggesting that not wearing dentures at night can worsen sleep quality and lead to severe sleep disturbance in edentate elders, there are also studies that have suggested the opposite. The current controversy does not permit clinicians to engage in evidence-based clinical decision-making. To enable development of clinical practice guidelines, solid evidence is required. This proposed randomized trial represents the logical next step of the clinical investigations conducted by our multidisciplinary expert team of oral health and sleep researchers from the University of Montreal, McGill University, University of British Colombia, and Laval University. Our pilot data suggest that edentate elders who wear dentures at night experience more daytime sleepiness than those who do not. Furthermore, we found that the nocturnal use of dentures may increase the risk of apneic events in seniors affected by mild sleep disturbance.

OBJECTIVES

The primary objective of this study is to test whether nocturnal denture wear has an effect on sleep quality and daytime sleepiness of edentate elders with moderate to severe sleep apnea. Our secondary objective is to test whether nocturnal denture wear affects on the oral-health-related quality of life of edentate elders with moderate to severe sleep apnea. . The third objective is to identify moderators of effect of nocturnal denture wear so as to determine patient subgroups where the intervention is more efficacious.

METHODS

We will carry out a single-blind randomized cross-over clinical trial, into which 70 edentate elders will be enrolled. Study participants will be assigned to wear and not wear their denture in alternate orders for two periods of 30 days. The primary outcome will be sleep quality (as measured by the apnea-hypopnea index). The secondary outcomes will be daytime sleepiness and oral health-related quality of life. Outcome assessments will be carried out with portable polysomnography, the Epworth Sleepiness Scale, and an oral health-related quality of life questionnaire. Explanatory variables will include socio-demographic factors, medical, and anthropometric (weight, height) variables, oropharyngeal morphology, oral and prosthesis characteristics, as well as perceived general health quality of life. These characteristics will be assessed by clinical examination, 3D imaging (Cone Beam Computed Tomography) of the cranio-facial structure, as well as validated questionnaires. Assessments will be done at baseline and at the end of each of the 30-day intervention periods. Linear mixed-effects regression models for repeated measures will be fitted to test the study hypotheses. The main analyses will be based on the intention-to-treat principle. To assess the robustness of the findings to potential incomplete adherence, sensitivity analyses will be conducted while applying the per-protocol principle.

SIGNIFICANCE

Our findings will have important clinical implications and will help to resolve the current uncertainty about the effects of nocturnal wearing of dentures in the edentate elderly population. This practice-relevant evidence could enable the development of preventive approaches to improve sleep quality of the older population and, thereby, improve their well-being and quality of life. This evidence will be shared with the Canadian Dental Association, the Canadian and the American Academy of Dental Sleep Medicine, and the Canadian Sleep Society to assist these agencies in producing practice guidelines for primary care providers, dentists, and sleep medicine specialists involved in the care of edentate elders.

ELIGIBILITY:
Inclusion Criteria:

* be aged 65 years or older; have worn a complete set of removable dentures in the last year AND not have worn a denture during sleep in the last 12 months;
* have an AHI ≥ 10 at screening
* have an adequate understanding of written and spoken English or French;
* be able to understand and respond to the questionnaires used in the study;
* agree to follow the research study instructions;
* agree to maximally adhere to the allocated sequence of interventions;
* consume no alcohol and not work late at night on the day before polysomnography.

Exclusion Criteria:

* have an AHI < 10;
* have any severe cardiologic, neurologic, psychological, or psychiatric condition, respiratory disease, acute airway infection or any other health condition that jeopardizes sleep;
* have a score of 24 or less on the mini-mental state evaluation;
* regularly consume more than 2 alcoholic beverages per day for females and 3 for males;
* are taking medication or any illicit drug that will affect sleep architecture or respiratory muscle activity (i.e., hypnotics, psychostimulants, anticonvulsant, or antipsychotics);
* are on regular continuous positive airway pressure therapy or nocturnal supplemental oxygen;
* have sleepiness deemed to be unsafe and requiring urgent treatment;
* feel that the trial would negatively influence their private life.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-04; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 30 days
  Sleep quality is measured by the AHI. The AHI index will be measured by use of diagnostic portable polysomnography.

SECONDARY OUTCOMES:
Daytime sleepiness | 30 days
  The Sleepiness Scale (ESS) will be used to assess perceived daytime sleepiness. Participants will be asked to rate their chance of dozing in eight different sedentary situations.
Oral health related quality of life | 30 days
  Oral health related quality of life will be measured by means of the oral health impact profile (OHIP-20). This instrument is a disease-specific measure of people's perceptions of their physical, psychological,and social impacts of oral health on their quality of life.

OTHER OUTCOMES:
Explanatory variables | Baseline
  These include socio-demographic, medical, and anthropometric (weight, height) variables, oropharyngeal morphology (measured by a 3-dimensional imaging system, CBCT, NewTom 5G CBCT, QR S.r.l.-Verona, Italy), edentulism-associated variables, as well as perceived general health. Perceived general health will be assessed by the use of the Short Form-36 (SF-36).

CONTACTS AND LOCATIONS:
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen H, Emami E, Kauffmann C, Rompre P, Almeida F, Schmittbuhl M, van der Stelt P, Ge S, Lavigne G, Huynh N. Airway Phenotypes and Nocturnal Wearing of Dentures in Elders with Sleep Apnea. J Dent Res. 2023 Mar;102(3):263-269. doi: 10.1177/00220345221133278. Epub 2022 Nov 4. PMID 36333889
- [Derived] Chen H, Elham E, Li Y, Ge S, Schmittbuhl M, Lavigne G, van der Stelt PF, Huynh N. Comparison of anatomic and aerodynamic characteristics of the upper airway among edentulous mild, moderate, and severe obstructive sleep apnea in older adults. J Clin Sleep Med. 2022 Mar 1;18(3):759-768. doi: 10.5664/jcsm.9716. PMID 34636319
- [Derived] Emami E, Lavigne G, Feine JS, Karp I, Rompre PH, Almeida FR, Huynh NT. Effects of nocturnal wearing of dentures on the quality of sleep and oral-health-related quality in edentate elders with untreated sleep apnea: a randomized cross-over trial. Sleep. 2021 Oct 11;44(10):zsab101. doi: 10.1093/sleep/zsab101. PMID 33955479
- [Derived] Emami E, Nguyen PT, Almeida FR, Feine JS, Karp I, Lavigne G, Huynh N. The effect of nocturnal wear of complete dentures on sleep and oral health related quality of life: study protocol for a randomized controlled trial. Trials. 2014 Sep 13;15:358. doi: 10.1186/1745-6215-15-358. PMID 25218696